CLINICAL TRIAL: NCT06117891
Title: An Observational Study in Patients With Unresectable Hepatocellular Carcinoma (uHCC) Following Treatment With Atezolizumab Plus Bevacizumab (AB) or With Another Approved Immuno-oncology Immune Checkpoint Inhibitor Combination in First-line
Brief Title: An Observational Study to Learn More About How Well a Treatment Works When Given After Treatment With Atezolizumab and Bevacizumab or Another Similar Combination of Drugs in Adults With Liver Cancer That Cannot be Treated With Surgery
Acronym: REFINE-IO
Status: Recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22453
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Unresectable Hepatocellular Carcinoma
Keywords: uHCC; systemic treatment; real-world data; prospective
MeSH Terms: interventions — atezolizumab; Bevacizumab; durvalumab; tremelimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment: Patients with a diagnosis of uHCC treated with first-line AB or another approved 1L-IO combo and in whom a decision to treat with a second-line of systemic therapy has been made by the treating physician at the time of study enrollment
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: Durvalumab; Drug: Tremelimumab,

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab combined with Bevacizumab, immune checkpoint inhibitors combination.
Drug: Bevacizumab — Atezolizumab combined with Bevacizumab, immune checkpoint inhibitors combination.
Drug: Durvalumab — Durvalumab combined with Tremelimumab, another immuno-oncology (IO) checkpoint inhibitors combination.
Drug: Tremelimumab, — Durvalumab combined with Tremelimumab, another immuno-oncology (IO) checkpoint inhibitors combination.

SUMMARY:
This is an observational study in which only data will be collected from adults with unresectable hepatocellular carcinoma. These adults should be prescribed a different treatment after treatment with atezolizumab and bevacizumab, or another similar combination of drugs, by their doctors.

Unresectable hepatocellular carcinoma (uHCC) is a type of liver cancer that cannot be treated with surgery.

In the past, sorafenib was the only approved first-line anti-cancer drug for people with uHCC. Regorafenib and other drugs were approved as second-line treatments for uHCC if a person could not take sorafenib or it stopped working for them.

Lately, another first-line (1L) treatment called immuno-oncology (IO) immune checkpoint inhibitor combination (1L-IO combo), like atezolizumab with bevacizumab (AB), has become the preferred choice of treatment. This is because of the meaningful impact on patient survival. 1L-IO combo are drugs that help the body's defense system recognize and kill cancer cells.

Since the other treatments were previously approved for use following sorafenib, the best order to take these treatments in following an 1L-IO combo is unknown.

To better understand and determine this order, more knowledge is needed about how well different treatments work in participants with uHCC who have been treated with AB or another 1L-IO combo.

The main purpose of this study is to learn more about how well different treatments work when given after first-line treatment with AB or another approved 1L-IO combo. To do this, researchers will collect data on how long the participants live (also called overall survival) from the start of any treatment given after the first-line treatment.

In addition, researchers will also collect the following information to learn more about the participants who will be given a different treatment after the 1L-IO combo:

* characteristics including age, sex, and race, and signs and symptoms of the participants over the duration of their first-line treatment
* the length of time from the first to the last dose (also called duration of therapy) of the treatments given after the 1L-IO combo
* the length of time until a participant's cancer worsens, or they die (also called progression free survival) from the start of the treatments given after the 1L-IO combo
* the number of participants whose tumor completely disappears or shrinks (also called overall tumor response) after taking the treatments given after the 1L-IO combo
* the sequence of treatments given after the 1L-IO combo Data will be collected from September 2023 to December 2026 and cover a period of around 3 years. The data will be collected using medical records or by interviewing the participants during their routine visits to the doctor.

Researchers will observe participants from the start of the treatment given after the 1L-IO combo until the end of their participation in the study.

In this study, only data from routine care will be collected. No visits or tests are required as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, ≥ 18 years of age on the day of signing informed consent.
* Confirmed diagnosis of uHCC, treated in a first-line setting with AB or another approved 1L-IO combo therapy.
* Decision to initiate treatment with a second-line systemic treatment was made as per investigator's routine treatment practice prior to study enrollment.
* Signed informed consent or (for patients under legal age) signed informed assent by the patient (where applicable) and signed informed consent by parents / legal guardian.
* No participation in an investigational program with interventions outside of routine clinical practice.

Exclusion Criteria:

- Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of uHCC treated with first-line AB or another approved 1L-IO combo and in whom a decision to treat with a second-line of systemic therapy has been made by the treating physician. The investigator or a delegate at these centers collects historic data (demographic and clinical characteristics) from medical records if available. The investigator or a delegate collects treatment-related data during visits that take place in routine practice.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2026-11-27 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Approximately 36 months
  OS is defined as the time (days) from start of second-line systemic treatment to the date of death, due to any cause. Patients alive or lost to follow-up will be censored at their last date of follow-up.

SECONDARY OUTCOMES:
Discriptive analysis of demographic characteristics | At baseline before the first drug administration of second-line systemic treatment
Discriptive analysis of clinical characteristics | At baseline before the first drug administration of second-line systemic treatment
Duration of therapy (DoT) | Approximately 36 months
  DoT in second-line setting will be calculated as the time (days) from the date of initiation of the second -line systemic treatment to the stop of this treatment regimen or to last date of follow-up, if treatment was ongoing on that date.
Progression-free survival (PFS) | Approximately 36 months
  PFS is defined as the time (days) from the date of initiation of systemic treatment to the earliest date of first observed disease progression (radiological or clinical) or death due to any cause.
Best overall response rate (ORR) | Approximately 36 months
  ORR will be defined according to investigator-assessed data according to local standard.
Treatment sequences post first-line AB or other IO combinations | Approximately 36 months

CONTACTS AND LOCATIONS:
Locations (20):
- United States (6):
  - Mercy Medical Center - Medline Healthcare Services LLC, Baltimore, Maryland
  - University of Michigan Health System, Ann Arbor, Michigan
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - University Of Cincinnati Division Of Hematology Oncology - UC Health System, Cincinnati, Ohio
  - Corporal Michael J Crescenz Department Of Veterans Affairs Medical Center, Philadelphia, Pennsylvania
  - Einstein Medical Center, Philadelphia, Pennsylvania
- Many Locations, Multiple Locations, Argentina
- Many Locations, Multiple Locations, Brazil
- Many Locations, Multiple Locations, China
- Many Locations, Multiple Locations, Colombia
- Many Locations, Multiple Locations, France
- Many Locations, Multiple Locations, Greece
- Many Locations, Multiple Locations, Italy
- Many Locations, Multiple Locations, Mexico
- Many Locations, Multiple Locations, Saudi Arabia
- Many Locations, Multiple Locations, South Korea
- Many Locations, Multiple Locations, Spain
- Many Locations, Multiple Locations, Taiwan
- Many Locations, Multiple Locations, Thailand
- Many Locations, Multiple Locations, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.